CLINICAL TRIAL: NCT07171840
Title: Effectiveness of Intra-articular Oxygen-ozone Injections and Splinting for the Treatment of Thumb Osteoarthritis: a Randomized Controlled Clinical Trial
Brief Title: Effectiveness of Intra-articular Oxygen-ozone Injections and Splinting for the Treatment of Thumb Osteoarthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Cristiano Sconza, Principal Investigator, Humanitas Clinical and Research Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OZTHUMB
Record Dates: First submitted 2025-09-06; First posted 2025-09-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Thumb Osteoarthritis
Keywords: oxygen-ozone; thumb splint; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone plus thumb splint (Experimental): Participant will receive an intraarticular injection of oxygen-ozone, once a week for two weeks. During procedure a clear ultrasound image is to be taken to document needle placement in the synovial space. After that, a physiotherapist will create two personalized thermoplastic splints for every patient for the stabilizing of the TMJ (one for the day that has a functional aim and one for the night with the objective of TMJ rest). The two splints will be used for 2 months.
  Interventions: Drug: 10 cc of oxygen-ozone plus thumb splint
- only thumb splint (Active Comparator): A physiotherapist will create two personalized thermoplastic splints for every patient for the stabilizing of the TMJ (one for the day that has a functional aim and one for the night with the objective of TMJ rest). The two splints will be used for 2 months.
  Interventions: Device: thumb splint

INTERVENTIONS:
Drug: 10 cc of oxygen-ozone plus thumb splint — Oxygene-Ozone therapy plus splint therapy
  Arms: ozone plus thumb splint
Device: thumb splint — thermoplastic splint
  Arms: only thumb splint

SUMMARY:
Osteoarthritis of trapezio-metacarpal joint (TMJ) most commonly occurs in women over 50 years old, often bilateral and it is a disabling condition presenting with pain at base of the thumb, swelling, instability, deformity and impairment of hand function with limitation in gripping and pinching objects. There are several surgical treatment options for TMJO as well as many conservative treatments such as splinting, thumb strengthening exercises, anti-inflammatory drugs and intra-articular injections. There are no currently approved TMJO treatments capable of slowing OA-related structural progression, so the main goals of the conservative treatment are to provide symptomatic relief, improve joint function, and delay surgical intervention. In recent years, the interest in the use of ozone is in constant increase especially because of the biological properties of inducing analgesia, anti-inflammatory, and antioxidant effects. Some articles have reported promising results on the effectiveness of oxygen-ozone, but the evidence is low. So, the aim of this study is to evaluate the effectiveness of intra-articular oxygen-ozone therapy (OOT) combined with thumb splint and compare it with only the splint therapy.

DETAILED DESCRIPTION:
Osteoarthritis is a degenerative condition that causes pain, impaired function and affects daily activities. In osteoarthritis, there is the destruction of cartilage and subchondral bone, with the consequent narrowing of articular space. Several factors have been associated with the development of degenerative changes in the carpometacarpal joint (CMCJ), including increased thumb base joint laxity and greater grip strength. Trapezio-metacarpal joint (TMJ) is a disabling condition presenting with pain at base of the thumb, swelling, instability, deformity and limitation of hand function. The patient with symptomatic TMJO in its initial stages is usually treated conservatively before surgical intervention: one of the main actions of intra-articular treatments, ranging from corticosteroids to hyaluronic acid and biologic products is to reduce inflammatory distress within the joint; injection treatments are usually used alone or in combination with thumb splint in a multimodal rehabilitation approach.

In recent years, there has been a growing interest in the effects of ozone because intra-articular administration of an adequate mixture of oxygen-ozone is supposed to reduce pain, to have protective immunomodulatory effects on cartilage, and to reduce oxidative stress, thus potentially representing an alternative to other injective methods. However, is still unclear what best therapeutic protocol is in terms of ozone concentration, volume to be injected, number of injections and time between injections.

This study will compare the efficacy of OOT injection plus thumb splint to only joint splint in patients with painful unilateral thumb OA who have been unable to achieve satisfactory pain relief with previous conservative OA treatment (e.g. physical therapy, simple analgesics). This will be done using a randomized controlled trial with study subjects receiving a cycle of two injection of OOT plus thumb splint. The primary study objective is to determine whether two injections of OO and thumb splint are superior to the use of only the joint splinting in reducing pain and this is measured by the improvement in DASH score from baseline. Secondary objectives of this study are improvement in VAS Pain, Grip Strength Function and Tip Pinch Function.

During screening, potential subjects who provide informed consent will be assessed for eligibility. Screening will consist in checking the presence of inclusion and exclusion criteria, including symptomatic OA in one thumb joint from 3 months and a thumb joint radiograph showing an Eaton and Litter grade of 1 to 3 and an absence of severe osteoarthritis. Subjects will also provide demographic and medication use information. Baseline X-ray will be collected.

ELIGIBILITY:
Exclusion Criteria:

1. Presence of clinically observed active infection or severe inflammation in the index trapezio-metacarpal joint or skin disease/breakdown or infection in the area of the planned injection site of the index thumb joint.
2. Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; Human Immunodeficiency Virus (HIV), viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis.
3. Diagnosed with leukaemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment.
4. Disease of cervical spine, shoulder or other upper extremity joints judged by the investigator to be contributing to the pain in the index thumb joint (e.g. radiculopathy, De Quervain S., etc.).
5. Untreated symptomatic injury of the index hand (e.g., acute traumatic injury, tendinopathy, nerve lesion).
6. Presence of surgical hardware or other foreign body intended to treat arthritis or cartilage-related pathology in the index thumb joint.
7. Presence of venous or lymphatic stasis in the index arm.
8. Orally administered systemic steroid use within 2 weeks prior to screening
9. Planned/anticipated surgery of the index hand during the study period.
10. Major surgery of the index hand within 12 months prior to screening.
11. Minor surgery (e.g. arthroscopy) of the index hand within 6 months prior to screening
12. Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening, which, in the opinion of the investigator, could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study injection.
13. Pregnant or nursing mothers or women planning to become pregnant during the time they will be participating in the study.
14. Previously documented failed treatment with OOT or splint
15. Known drug or alcohol dependence currently or within the last year.
16. Use of any investigational drug or device within 30 days prior to screening.
17. Use of any investigational biologics within 60 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-23 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) | 1, 3, 6 months
  Assessment of the patient's disability; 38 questions, score range 0-100. Higher scores indicate greater severity of disability.

SECONDARY OUTCOMES:
Visual Analogic Scale (VAS) | 1, 3, 6 months
  Assessment of pain. Score range 0-10. Higher scores indicate worse pain.
Grip strength test | 1,3,6 months
  Assessment of force. It tests muscles responsible for flexion of the metatarsals and phalanges. Changes in force are recorded by the use of a dynamometer
Tip pinch strength test | 1, 3, 6 months
  Assessment of force. It tests muscles responsible for flexion of the fingers and adduction of the thumb. Changes in force are recorded by the use of a dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-09-23): https://cdn.clinicaltrials.gov/large-docs/40/NCT07171840/Prot_SAP_000.pdf